CLINICAL TRIAL: NCT02485210
Title: Evaluation of the Effectiveness of Photodynamic Therapy as a Supporting for Endodontic Treatment of Deciduous Teeth
Brief Title: Effectiveness of Photodynamic Therapy for Endodontic Treatment of Deciduous Teeth
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Nove de Julho (Other)
Responsible Party: Principal Investigator, Sandra Kalil Bussadori, Dr., University of Nove de Julho
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 832.657
Record Dates: First submitted 2015-06-09; First posted 2015-06-30 (Estimated); Last update posted 2017-05-08 (Actual); Status verified 2017-05

CONDITIONS: Tooth, Nonvital
Keywords: photodynamic therapy , Endodontic treatment
MeSH Terms: conditions — Tooth, Nonvital | interventions — Endodontics

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Covencional treatment (Active Comparator): Convencional endodontic treatment for deciduous teeth, with Surgical chemical preparation with series of Kerr files appropriate for each case, using initial file and an additional two files of larger size, with irrigation and aspiration with 1% sodium hypochlorite (Milton's solution) and endo PTC (Fórmula & Ação) with each change of file.
  Filling of root canals with calcium hydroxide (Ultra-cal, Ultradent, Brazil); base of thin gutta-percha and filling with glass ionomer cement; restorative treatment performed in subsequent session.
  Interventions: Procedure: Endodontic treatment
- Photodynamic therapy (Experimental): Endodontic Treatment with photodynamic terapy Irrigation of the root canal system Insertion of sterile paper cone immersed in Chimiolux® methylene blue for three minutes; administration of wireless Therapy XT EC laser device (DMC - São Carlos, Brazil) after removal of cone; energy density: 4 J/cm², power: 100 mw; wavelength: 660 nm; exposure time: 40 seconds Filling of root canals with calcium hydroxide (Ultra-cal, Ultradent, Brazil); base of thin gutta-percha and filling with glass ionomer cement; restorative treatment performed in subsequent session
  Interventions: Procedure: Endodontic treatment

INTERVENTIONS:
Procedure: Endodontic treatment — It will be done the endodontic treatment using the photosynamic therapy for decontamination of the root chanel.

SUMMARY:
The elimination of pathogenic microorganisms from the root canal system is one of the main points in order to have success in endodontic treatment. The objective of this study is to perform a randomized controlled clinical trial to compare the effectiveness of success in endodontic treatment of primary teeth when combined with photodynamic therapy. Will be selected 30 primary teeth of children aged between 3 and 6 years. The teeth will be divided into two groups: group I control, which will be applied the conventional endodontic treatment and group II to be held endodontic treatment with application of photodynamic therapy. In both groups will be made microbiological evaluations before and after endodontic treatment and clinical and radiographic evaluations will be conducted in the day, 1 month, 3 months and 6 months after treatment comparing the treatment performed in both groups.

DETAILED DESCRIPTION:
Interventions All treatment procedures will be performed by a single, duly trained operator. Group I (control) - conventional endodontic treatment

1. Prophylaxis with pumice stone and water and antisepsis of region with 0.12% solution of chlorhexidine using moistened gauze
2. Anesthesia
3. Absolute isolation, if possible; in cases of considerable loss of remaining tooth, relative isolation using cotton rolls
4. Opening of crown with spherical diamond tip burs (bur size compatible with tooth) (KG Sorensen - Indústria e Comércio, SP, Brazil) and high speed Z endodontic drill under water and air refrigeration
5. Millimeter measurement of root canal to 1 mm short of radiographic apex
6. Insertion of three sterile paper cones with diameter compatible with canal for 30 seconds for initial collection of bacterial sample and immediate placement into brain heart infusion broth
7. Surgical chemical preparation with series of Kerr files appropriate for each case, using initial file and an additional two files of larger size, with irrigation and aspiration with 1% sodium hypochlorite (Milton's solution) and endo PTC (Fórmula & Ação) with each change of file
8. Insertion of three sterile paper cones for 30 seconds for second collection of bacterial sample and immediate placement into brain heart infusion broth
9. Filling of root canals with calcium hydroxide (Ultra-cal, Ultradent, Brazil); base of thin gutta-percha and filling with glass ionomer cement; restorative treatment performed in subsequent session

Group II - Conventional endodontic treatment + PDT

1. Prophylaxis with pumice stone and water and antisepsis of region with 0.12% solution of chlorhexidine using moistened gauze
2. Anesthesia
3. Absolute isolation, if possible; in cases of considerable loss of remaining tooth, relative isolation using cotton rolls
4. Opening of crown with spherical diamond tip burs (bur size compatible with tooth) (KG Sorensen - Indústria e Comércio, SP, Brazil) and high speed Z endodontic drill under water and air refrigeration
5. Millimeter measurement of root canal to 1 mm short of radiographic apex
6. Insertion of three sterile paper cones with diameter compatible with canal for 30 seconds for initial collection of bacterial sample and immediate placement into brain heart infusion broth
7. Insertion of sterile paper cone immersed in Chimiolux® methylene blue for three minutes; administration of wireless Therapy XT EC laser device (DMC - São Carlos, Brazil) after removal of cone; energy density: 4 J/cm², power: 100 mw; wavelength: 660 nm; exposure time: 40 seconds
8. Root canal irrigated with sterile saline solution and insertion of three sterile paper cones for 30 seconds for second collection of bacterial sample and immediate placement in brain heart infusion broth
9. Filling of root canals with calcium hydroxide (Ultra-cal, Ultradent, Brazil); base of thin gutta-percha and filling with glass ionomer cement; restorative treatment performed in subsequent session

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 3 to 6 years old with at least one anterior deciduous tooth with irreversible pulpitis or pulp necrosis in a position to be restored and at least 2/3 of the remaining root.
* Healthy patients and who did not antibiotic treatment in the previous three months.

Exclusion Criteria:

* Patients in poor health, with primary teeth with large root loss (+ 2/3 root), which has no internal pathological resorption, reconstruction is not possible, cases of retreatment and crypt involvement.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Estimated)
Dates: Start 2017-04-29 (Actual); Primary Completion 2017-10 (Estimated); Study Completion 2018-04 (Estimated)

PRIMARY OUTCOMES:
Clinical evaluation. | 6 months
  If the teeth doesn´t has any sympton like pain, fistula etc...

SECONDARY OUTCOMES:
Radiographic evaluation | 6 mounth
  Periapical lesion (Yes or No).
Microbiological evaluation | Before and after the treatment (same day)
  UFC/ml before and after treatment

CONTACTS AND LOCATIONS:
Overall Officials: Sandra Bussadori, PhD, Principal Investigator — University of Nove de Julho
Locations (1):
- University of Nove de Julho, São Paulo, Brazil

REFERENCES:
- [Derived] da Mota AC, Goncalves ML, Bortoletto C, Olivan SR, Salgueiro M, Godoy C, Altavista OM, Pinto MM, Horliana AC, Motta LJ, Bussadori SK. Evaluation of the effectiveness of photodynamic therapy for the endodontic treatment of primary teeth: study protocol for a randomized controlled clinical trial. Trials. 2015 Dec 3;16:551. doi: 10.1186/s13063-015-1086-2. PMID 26635011